CLINICAL TRIAL: NCT05864547
Title: Predisposing Factors for Post-stroke Epilepsy
Acronym: PRESTEP
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 527577
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Post Stroke Epilepsy; Stroke; Epilepsy; Seizures
Keywords: Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Disorders; Vascular Diseases
MeSH Terms: conditions — Stroke; Epilepsy; Seizures; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months

GROUPS / COHORTS (2):
- Stroke patients: Patients with first time stroke admitted to the stroke unit, St. Olavs hospital, Trondheim, Norway. The planned cohort size is 15-20 patients.
- Healthy controls: Age and gender matched healthy volunteers without previous stroke. The same number of healthy controls as recruited patients will be recruited through ads in the local newspaper.

SUMMARY:
The goal of this observational study is to learn about epilepsy after a stroke (post-stroke epilepsy). The main questions it aims to answer are:

* What make some patients develop epilepsy after a stroke?
* Does sleep have an impact on the development of post-stroke epilepsy?

Participants will undergo:

* Electroencephalography (EEG)
* Magnetic resonance imaging (MRI)
* Polysomnography (only patients)

Blood tests will also be taken. The patient group will be compared to the healthy controls. Researchers will also look into medical records of stroke patients hospitalized at St. Olavs hospital and collect relevant information.

DETAILED DESCRIPTION:
This study aims to study risk factors and clinical factors which might contribute to the development of post-stroke epilepsy. Researchers will look at the volume and size of the stroke-induced brain lesions and analyze inflammation markers. Patients and controls will undergo EEG and MRI. The correlations between sleep and epilepsy after a stroke will also be investigated through polysomnography. Relevant information about for instance age, comorbidities and NIHSS will be collected. Researchers will also collect relevant information from medical records of stroke patients hospitalized at St. Olavs hospital.

ELIGIBILITY:
Inclusion Criteria:

* First time stroke patients with capacity to consent, admitted to the stroke unit at St. Olavs hospital.
* Modified Rankin Scale (mRS) ≤ 2 before the stroke

Exclusion Criteria:

* Previous stroke or brain surgery
* Traumatic brain injuries
* Neurodegenerative diseases
* Brain tumors
* Epilepsy before the stroke
* Hydrocephalus
* Aphasia
* Serious psychiatric disorders
* MRI incompatibility and claustrophobia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First time stroke patients with capacity to consent and who can undergo MR imaging, admitted to the stroke unit at St. Olavs hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Post-stroke epilepsy | 6 months
  Minimum one documented case of post-stroke epilepsy after the stroke

SECONDARY OUTCOMES:
Acute symptomatic seizure | 14 days
  Minimum one documented case of acute symptomatic seizure with epileptogenic activity recorded with EEG

CONTACTS AND LOCATIONS:
Overall Officials: Axel Sandvig, PhD prof, Principal Investigator — Norwegian Science and Technology University
Locations (1):
- St. Olavs Hospital Stroke Unit, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bentes C, Martins H, Peralta AR, Morgado C, Casimiro C, Franco AC, Fonseca AC, Geraldes R, Canhao P, Pinho E Melo T, Paiva T, Ferro JM. Early EEG predicts poststroke epilepsy. Epilepsia Open. 2018 Mar 7;3(2):203-212. doi: 10.1002/epi4.12103. eCollection 2018 Jun. PMID 29881799
- [Background] Pitkanen A, Roivainen R, Lukasiuk K. Development of epilepsy after ischaemic stroke. Lancet Neurol. 2016 Feb;15(2):185-197. doi: 10.1016/S1474-4422(15)00248-3. Epub 2015 Nov 17. PMID 26597090
- [Background] Wang G, Jia H, Chen C, Lang S, Liu X, Xia C, Sun Y, Zhang J. Analysis of risk factors for first seizure after stroke in Chinese patients. Biomed Res Int. 2013;2013:702871. doi: 10.1155/2013/702871. Epub 2013 Nov 2. PMID 24298553
- [Background] Duss SB, Seiler A, Schmidt MH, Pace M, Adamantidis A, Muri RM, Bassetti CL. The role of sleep in recovery following ischemic stroke: A review of human and animal data. Neurobiol Sleep Circadian Rhythms. 2016 Nov 29;2:94-105. doi: 10.1016/j.nbscr.2016.11.003. eCollection 2017 Jan. PMID 31236498
- [Background] Zollner JP, Schmitt FC, Rosenow F, Kohlhase K, Seiler A, Strzelczyk A, Stefan H. Seizures and epilepsy in patients with ischaemic stroke. Neurol Res Pract. 2021 Dec 6;3(1):63. doi: 10.1186/s42466-021-00161-w. PMID 34865660
- [Background] Arntz RM, Rutten-Jacobs LC, Maaijwee NA, Schoonderwaldt HC, Dorresteijn LD, van Dijk EJ, de Leeuw FE. Poststroke Epilepsy Is Associated With a High Mortality After a Stroke at Young Age: Follow-Up of Transient Ischemic Attack and Stroke Patients and Unelucidated Risk Factor Evaluation Study. Stroke. 2015 Aug;46(8):2309-11. doi: 10.1161/STROKEAHA.115.010115. Epub 2015 Jul 2. PMID 26138118
- [Background] Hassani M, Cooray G, Sveinsson O, Cooray C. Post-stroke epilepsy in an ischemic stroke cohort-Incidence and diagnosis. Acta Neurol Scand. 2020 Feb;141(2):141-147. doi: 10.1111/ane.13174. Epub 2019 Oct 22. PMID 31580473
- [Background] Jungehulsing GJ, Heuschmann PU, Holtkamp M, Schwab S, Kolominsky-Rabas PL. Incidence and predictors of post-stroke epilepsy. Acta Neurol Scand. 2013 Jun;127(6):427-30. doi: 10.1111/ane.12070. Epub 2013 Feb 7. PMID 23398544
- [Background] Zollner JP, Misselwitz B, Kaps M, Stein M, Konczalla J, Roth C, Krakow K, Steinmetz H, Rosenow F, Strzelczyk A. National Institutes of Health Stroke Scale (NIHSS) on admission predicts acute symptomatic seizure risk in ischemic stroke: a population-based study involving 135,117 cases. Sci Rep. 2020 Mar 2;10(1):3779. doi: 10.1038/s41598-020-60628-9. PMID 32123219
- [Background] De Reuck J, Goethals M, Claeys I, Van Maele G, De Clerck M. EEG findings after a cerebral territorial infarct in patients who develop early- and late-onset seizures. Eur Neurol. 2006;55(4):209-13. doi: 10.1159/000093871. Epub 2006 Jun 13. PMID 16772712